CLINICAL TRIAL: NCT03273335
Title: Investigating NeuroinflammaTion UnderlyIng Postoperative Brain Connectivity Changes, POCD, Delirium in Older Adults
Acronym: INTUIT
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00083288; 1K76AG057022 (NIH)
Record Dates: First submitted 2017-09-03; First posted 2017-09-06 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CSF, Blood/Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Surgical patients: Surgical patients will undergo CSF biomarker assays, cognitive testing and fMRI scans.
  Interventions: Device: Millipore biomarker assay plate

INTERVENTIONS:
Device: Millipore biomarker assay plate — Millipore biomarker assay plate CSF cytokine assays as well as CSF flow cytometry

SUMMARY:
(From NIH reporter) Each year >16 million older Americans undergo anesthesia and surgery, and up to 40% of these patients develop postoperative cognitive dysfunction (POCD), a syndrome of postoperative thinking and memory deficits. Although distinct from delirium, POCD (like delirium) is associated with decreased quality of life, long term cognitive decline, early retirement, increased mortality, and a possible increased risk for developing dementia such as Alzheimer's disease. Understanding the etiology of POCD will likely help promote strategies to treat and/or prevent it. A dominant theory holds that brain inflammation causes POCD, but little work has directly tested this theory in humans. The preliminary data of this team strongly suggest that there is significant postoperative neuro-inflammation in older adults who develop POCD. In this K76 award, the investigators will prospectively obtain pre- and post-operative cognitive testing, fMRI imaging and CSF samples in 200 surgical patients over age 65. This will allow the investigators to evaluate the role of specific neuro-inflammatory processes in POCD and its underlying brain connectivity changes.

DETAILED DESCRIPTION:
Each year >16 million older Americans undergo anesthesia and surgery, and up to 40% of these patients develop postoperative cognitive dysfunction (POCD), a syndrome of postoperative thinking and memory deficits. Although distinct from delirium, POCD (like delirium) is associated with decreased quality of life, long term cognitive decline, early retirement, increased mortality, and a possible increased risk for developing dementia such as Alzheimer's disease. Understanding the etiology of POCD will likely help promote strategies to treat and/or prevent it. A dominant theory holds that brain inflammation causes POCD, but little work has directly tested this theory in humans. The preliminary data of this team strongly suggest that there is significant postoperative neuro-inflammation in older adults who develop POCD. In this K76 award, the investigators will prospectively obtain pre- and post-operative cognitive testing, fMRI imaging and CSF samples in 200 surgical patients over age 65. This will allow the investigators to evaluate the role of specific neuro-inflammatory processes in POCD and its underlying brain connectivity changes.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and above
* Having surgery scheduled to last > or = to 2 hours at Duke University Medical Center (ie Duke Hospital, Duke Medicine Pavilion, Duke Regional Hospital, Durham VA, Duke Raleigh Hospital)

Exclusion Criteria:

* Anticoagulants (per ASRA guidelines)
* Current use of chemotherapeutic agents with known cognitive effects.

Ages: 60 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients age 60 and above, as described above.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Correlation between Perioperative changes in CSF Monocytes and perioperative changes in cognition (continuous cognitive index change) | from before to 6 weeks after anesthesia/surgery
  as above

CONTACTS AND LOCATIONS:
Overall Officials: Miles Berger, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berger M, Murdoch DM, Staats JS, Chan C, Thomas JP, Garrigues GE, Browndyke JN, Cooter M, Quinones QJ, Mathew JP, Weinhold KJ; MADCO-PC Study Team. Flow Cytometry Characterization of Cerebrospinal Fluid Monocytes in Patients With Postoperative Cognitive Dysfunction: A Pilot Study. Anesth Analg. 2019 Nov;129(5):e150-e154. doi: 10.1213/ANE.0000000000004179. PMID 31085945